CLINICAL TRIAL: NCT02313740
Title: Prospective Cohort Study to Evaluate Safety and Immunogenicity of Butantan´s Fragmented, Inactivated Trivalent Influenza Vaccine in Healthy Adults and Elderly
Brief Title: Prospective Cohort Study to Evaluate Safety/Immunogenicity of Butantan Influenza Vaccine in Healthy Adults/Elderly
Status: Completed | Type: Observational
Sponsor: Butantan Institute (Other Government)
Responsible Party: Sponsor
Other Study IDs: FLU-04-IB
Record Dates: First submitted 2014-12-04; First posted 2014-12-10 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Influenza
Keywords: Influenza; Influenza Vaccines
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy adults group: Healthy adults aged 18 to 59 years Butantan Fragmented Inactivated Trivalent Influenza Vaccine
  Interventions: Biological: Butantan Fragmented Inactivated Trivalent Influenza Vaccine
- Elderly group: Elderly aged over than 60 years completed Butantan Fragmented Inactivated Trivalent Influenza Vaccine
  Interventions: Biological: Butantan Fragmented Inactivated Trivalent Influenza Vaccine

INTERVENTIONS:
Biological: Butantan Fragmented Inactivated Trivalent Influenza Vaccine — Subjects participating in the study are exposed to Butantan´s Fragmented Inactivated Trivalent Influenza Vaccine during vaccination campaign, and will have immunogenicity and safety related to the vaccine evaluated (observational study).

SUMMARY:
Prospective cohort study to evaluate safety and immunogenicity of the fragmented, inactivated trivalent Influenza vaccine produced at Butantan Institute in healthy adults and elderly. The study will include a total of 120 participants: 60 participants aged 18 to 59 years in the healthy adults group, and 60 participants aged older than 60 years in the elderly group.This study will evaluate the safety of one dose of the fragmented, inactivated trivalent Influenza vaccine in the first 3 days after vaccination, as well as its immunogenicity 21 days after vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults, male or female aged 18 to 59
* Elderly aged 60 years completed and above
* To be available to participate in the study throughout its duration (approximately 21 days)
* To have medical indication to be vaccinated against influenza
* To demonstrate intention to participate in the study, as documented by signature in the study´s informed consent form.

Exclusion Criteria:

* Evidence of active neurological, cardiac, pulmonary, hepatic or renal disease as clinical history and/or physical examination (except hypertension under control among the elderly)
* Compromised immune system diseases including: HIV, diabetes mellitus, cancer (except basal cell carcinoma) and autoimmune diseases
* Behavioral, cognitive or psychiatric disease that in the opinion of the principal investigator or his representative physician, affects the participant ability to understand and cooperate with all study protocol requirements
* Abusive usage of alcohol or drugs in the past 12 months that has caused medical, professional or family problems, indicated by clinical history
* Known systemic hypersensitivity to eggs or to any component of the vaccine
* History of severe adverse reaction after previous administration of an Influenza vaccine within 6 weeks following vaccination
* History of Guillain-Barre Syndrome or other demyelinating disease
* Diagnosis of asthma with a history of hospitalization in the last six months due to illness
* Suspected or confirmed fever in the 3 days prior to vaccination or axillary temperature greater than 37.8 ° C on the day of vaccination
* Use of corticosteroids (except topical or nasal) or other immunosuppressive drugs within 42 days before study initiation/baseline. It will be considered immunosuppressive dose of corticosteroids the equivalent to a dose ≥10 mg of prednisone per day for over 14 days
* Impaired coagulation due to chronic disease or due to use anticoagulant medication (warfarin or heparin) in the 7 days preceding vaccination
* Have received live virus vaccine within 28 days or killed virus vaccine in the last 14 days prior to vaccination, or have a scheduled immunization during the first 21 days after vaccination
* Have received influenza vaccine in the past 6 months;
* History of asplenia
* Have received blood products in the past 6 months, including transfusions or immunoglobulin, or scheduled administration of blood products or immunoglobulin for the first 21 days after vaccination
* have a counterindication for Influenza vaccination, including allergy to egg proteins
* Use of any investigational product within 42 days before vaccination;
* Any other condition that might put in risk the safety/rights of a potential participant or hurdle his/her compliance with this protocol in investigator's opinion or his representative physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Health adults with age between 18 and 59 years, as well as elderly over 60 years of age may participate in the study. To be included in the study, participants need to meet all inclusion criteria, and not fulfill any exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2015-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Vaccine Immunogenicity | 21 days
  Antibody response to each of the vaccine´s strains as measured by % seroconversion, increase in the geometric mean of hemagglutination-inhibition (HAI) titers and % seroprotection.
Vaccine safety assessed by unsolicited local and systemic adverse reactions up to 3 days post vaccination | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Alex R Precioso, MD, PhD, Study Director — Butantan Institute

REFERENCES:
- [Derived] Mondini G, Braga PE, Lopes MH, Sartori AMC, Miyaji KT, Infante V, Randi BA, Timenetsky MDCST, Ferreira JCOA, Sakita NK, Precioso AR. Prospective cohort studies to evaluate the safety and immunogenicity of the 2013, 2014, and 2015 seasonal influenza vaccines produced by Instituto Butantan. Rev Inst Med Trop Sao Paulo. 2018 Jul 30;60:e37. doi: 10.1590/S1678-9946201860037. PMID 30066805